CLINICAL TRIAL: NCT00856076
Title: Venous Thromboembolism and Intrauterine Fetal Death in Pregnancy - Epidemiology and Pathogenic Mechanisms
Brief Title: Venous Thromboembolism in Pregnancy Study
Acronym: VIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VIP-study
Record Dates: First submitted 2009-03-04; First posted 2009-03-05 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2009-03

CONDITIONS: Venous Thromboembolism; Intrauterine Fetal Death
Keywords: Venous thromboembolism; Intrauterine fetal death; Risk factor; Thrombophilia; Venous thromboembolism (in pregnancy)
MeSH Terms: conditions — Venous Thromboembolism; Stillbirth; Thrombophilia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, EDTA and citrated plasma, whole blood and processed DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- VTE case group 1/2: Women with first time venous thromboembolism in pregnancy. VTE data validated from medical records.
- VTE control group 1: All pregnancies of source population - clinical data from the Norwegian Birth Registry and the Norwegian Patient Registry.
- VTE control group 2: Randomly drawn from group 1 (using the Norwegian Birth Registry), but matched for time of delivery. Without history of venous thromboembolism, and with validated data from medical records.
- VTE case group 3: Subjects from VTE case group 1/2 invited to meet for investigation, donation of biological material and to answer a questionnaire.
- VTE control group 3: Subjects from VTE control group 2 invited to meet for investigation, donation of biological material and to answer a questionnaire.
- IUFD group 1: Women who have experienced IUFD - data verified from medical records.
- IUFD group 2: Subjects from IUFD group 2 invited to meet for investigation, donation of biological material and to answer a questionnaire.
- IUFD control group 1: All pregnancies of source population - clinical data from the Norwegian Birth Registry and the Norwegian Patient Registry.
- IUFD control group 2: Subjects from VTE control group 1/2 with validated data from medical records.
- IUFD control group 3: Subjects from VTE control group 3 invited to answer a disease specific questionnaire for IUFD.

SUMMARY:
The purpose of this study is to investigate clinical, biochemical and genetic risk factors for venous thromboembolism in pregnancy and pregnancy related vascular complications, and the long-term outcome of such complications including implications for quality of life.

DETAILED DESCRIPTION:
Background: Venous thromboembolism (VTE) in pregnancy is a serious, but rare condition. There is no epidemiological data on this patient group from Norway, and there is generally little literature on the immediate and long-term outcome after such pregnancies. Approximately 50% of the women with VTE in pregnancy have known thrombophilia. These women also carry a considerably increased risk for intrauterine fetal death (IUFD). In this project we want to identify new thrombophilias as risk factors for VTE and IUFD in pregnancy.

Aims:

Using a case-control design we will investigate the following issues:

* Risk factors for VTE in pregnancy and IUFD
* Association between thrombophilia, VTE, and other vascular pregnancy complications including IUFD
* Association between thrombophilia and IUFD
* Long term effects of VTE in pregnancy and IUFD on future health including quality of life
* Association between "single nucleotide polymorphisms" (SNP) in genes coding for specific coagulation-, fibrinolysis-, inflammatory, and other relevant proteins and their phenotypic expression
* Association between relevant phenotypes of coagulation, fibrinolysis, inflammation, and other relevant pathways and their risk of disease
* Association between the frequency of specific SNPs that codes for coagulation-, fibrinolysis-, inflammatory, and other relevant proteins and risk for VTE

Materials and Methods:

* 300 women with a history of VTE in their pregnancy and 150 women with IUFD will be identified by the Norwegian patient registry (NPR) and the Medical Birth Registry (MFR). The medical records of these patients will be checked. The epidemiological data will be collected with the help of questionnaires that the patients will fill out and blood samples will be collected. Blood samples will be analyzed with the aim to check for known coagulation factors and thrombophilias as well as new gene polymorphisms.
* 600 control women, from the maternity wards at Ullevål/Aker University Hospitals in the same time period, matched for age and ethnicity, will also answer questionnaires and donate blood samples. The medical records for these women will be checked.

Ethical problems: This study raises no new ethical problems. The study is based on voluntary participation from the invited and informed consent for all analyzes of biological test material. The study design, data procedures and storing of biological material, will use methods that assure the patients privacy at all levels.

The participants are invited to fill out a questionnaire concerning information of thrombosis in pregnancy and take one simple blood test. Women with symptoms of post thrombotic syndrome (PTS) will be offered a clinical examination of their lower extremities to verify the condition. The data will be de-identified and the individuals will not be able to be identify by other than those that have concession to the patient register established for this study.

Blood tests will be stored in a biobank at Ullevål University Hospital (UUS) established for this study, and will only be used for research related problems that have to do with this study.

Some patients could have a psychological reaction of the illness they experienced many years ago. The project leader or co-workers from the Hematology Department/Research Laboratory will handle this problem. These patients will be offered additional information on thrombosis in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* women with first-time objectively verified venous thromboembolism in pregnancy.
* women with history of intrauterine fetal death.

Exclusion Criteria:

* recurrent venous thromboembolism in pregnancy.
* non-validated venous thromboembolism in pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases: women with first-time validated venous thromboembolism in pregnancy or women who had experienced intrauterine fetal death, either all cases with validated data from medical records or cases meeting for blood sampling.
  Controls: women from the source population; either population based with data from the Norwegian Patient Registry or Norwegian Birth Registry, or hospital-based and randomly drawn from the source population and with validated data, or subset of the latter group meeting for blood sampling
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2023-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Per Morten Sandset, MD, PhD, Study Director — Oslo University Hospital Ullevål and University of Oslo
Locations (2):
- Norway (2):
  - Oslo University Hospital Ullevaal (formerly Ullevaal University Hospital), Oslo
  - Oslo University Hospital (formerly Ullevaal University Hospital), Oslo

REFERENCES:
- [Background] Bergrem A, Jacobsen EM, Skjeldestad FE, Jacobsen AF, Skogstad M, Sandset PM. The association of antiphospholipid antibodies with pregnancy-related first time venous thrombosis--a population-based case-control study. Thromb Res. 2010 May;125(5):e222-7. doi: 10.1016/j.thromres.2009.12.006. Epub 2010 Jan 6. PMID 20051285
- [Result] Jacobsen AF, Skjeldestad FE, Sandset PM. Incidence and risk patterns of venous thromboembolism in pregnancy and puerperium--a register-based case-control study. Am J Obstet Gynecol. 2008 Feb;198(2):233.e1-7. doi: 10.1016/j.ajog.2007.08.041. Epub 2007 Nov 12. PMID 17997389
- [Result] Jacobsen AF, Skjeldestad FE, Sandset PM. Ante- and postnatal risk factors of venous thrombosis: a hospital-based case-control study. J Thromb Haemost. 2008 Jun;6(6):905-12. doi: 10.1111/j.1538-7836.2008.02961.x. Epub 2008 Mar 21. PMID 18363820
- [Derived] Gravensteen IK, Helgadottir LB, Jacobsen EM, Radestad I, Sandset PM, Ekeberg O. Women's experiences in relation to stillbirth and risk factors for long-term post-traumatic stress symptoms: a retrospective study. BMJ Open. 2013 Oct 22;3(10):e003323. doi: 10.1136/bmjopen-2013-003323. PMID 24154514
- [Derived] Gravensteen IK, Helgadottir LB, Jacobsen EM, Sandset PM, Ekeberg O. Long-term impact of intrauterine fetal death on quality of life and depression: a case-control study. BMC Pregnancy Childbirth. 2012 Jun 7;12:43. doi: 10.1186/1471-2393-12-43. PMID 22676992
- [Derived] Jacobsen AF, Dahm A, Bergrem A, Jacobsen EM, Sandset PM. Risk of venous thrombosis in pregnancy among carriers of the factor V Leiden and the prothrombin gene G20210A polymorphisms. J Thromb Haemost. 2010 Nov;8(11):2443-9. doi: 10.1111/j.1538-7836.2010.04038.x. PMID 20735725